CLINICAL TRIAL: NCT02435797
Title: Effect of Early Administration of Intracoronary Nicorandil Via Thrombus Aspiration Catheter Device During Primary Percutaneous Coronary Intervention for the Patients of Acute ST Segment Elevation Myocardial Infarction
Brief Title: Effect of Nicorandil for the Patients of Acute ST Segment Elevation Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Feng Chunguang, Associate Professor, Xuzhou Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: W201416
Record Dates: First submitted 2015-04-23; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Heart Disease
Keywords: nicorandil; primary percutaneous coronary intervention; acute ST segment elevation myocardial infarction; thrombus aspiration
MeSH Terms: conditions — Coronary Disease; ST Elevation Myocardial Infarction | interventions — Nicorandil; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil (Active Comparator): Nicorandil for injection
  Interventions: Drug: Nicorandil
- normal saline (Placebo Comparator): normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Nicorandil — All patients received antiplatelet agents (aspirin, ticagrelor) and heparin.Diagnostic coronary angiography (CAG) was performed via the right (or left) femoral artery or radial artery using the Seldinger method.The guidewire was passed into the culprit lesion. Subjects in the NicorandilGroup were then given 2 mg intracoronary nicorandil through the lesions via thrombus aspiration catheter, and an additional intracoronary dose of 2 mg nicorandil before stent implantation. A minimum 5-min interval occurred between the first and second doses of nicorandil to reduce adverse effects.
  Arms: Nicorandil
Drug: normal saline — All patients received antiplatelet agents (aspirin, ticagrelor) and heparin.Diagnostic coronary angiography (CAG) was performed via the right (or left) femoral artery or radial artery using the Seldinger method.The guidewire was passed into the culprit lesion. Normal saline in the Placebo Group were then given 2 ml through the lesions via thrombus aspiration catheter,and an additional intracoronary dose of 2 ml before stent implantation. A minimum 5-min interval occurred between the first and second injection.
  Arms: normal saline

SUMMARY:
To evaluate whether nicorandil as an adjunctive therapy for acute myocardial infarction (AMI) reduces reperfusion injury.

DETAILED DESCRIPTION:
Reperfusion injury might occur in patients with acute ST segment elevation myocardial infarction undergoing the primary percutaneous coronary intervention(P-PCI),characterized by myocardial stunning, reperfusion-induced arrhythmia, microvascular dysfunction and myocardial cellular apoptosis, etc.

Nicorandil is an antianginal agent with a dual mechanism of action: nitrate and K+ATP channel opener. The nitrate action causes vasodilation of systemic veins and epicardial coronary arteries, while the adenosine triphosphate (ATP)-sensitive potassium channel opener action causes vasodilation of peripheral and coronary resistance arterioles. Nicorandil not only decreases preload and afterload but also increases coronary blood flow.

The study will compare the effectiveness between nicorandil and placebo of preventing the reperfusion injury and left ventricle remodeling in patients with acute ST segment elevation myocardial infarction undergoing the P-PCI.It is intended that before reperfusion injury ,nicorandil which was early used by intracoronary injection could prevent and release the microcirculatory spasm, release the coronary microvascular endothelial swelling,decrease embolism of atherosclerotic debris and thrombus formation.So,it could decrease the phenomenon of no-reflow/slow reflow,reperfusion-induced arrhythmia and worsening of chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST Segment Elevation Myocardial Infarction (ASTEMI) defined as typical chest pain lasting >30min within the previous 12 h, with a clear ST-segment elevation of >0.1millivolt(mV) in ≥2 contiguous electrocardiographic leads, and the value of troponin I(TNI) above the maximum peak in the normal range.
* Age20-80,All genders
* The first myocardial infarction, and there is no history of PCI therapy and coronary artery bypass grafting
* The infarct-related artery(IRA) is totally occlusive
* Blood pressure is higher than 90/60 millimeters of mercury（mmHg）
* The time from myocardial infarction onset to reach the hospital is less than 12 hs
* Successful interventional treatment, the residual stenosis of IRA is less than 30% ,
* TIMI flow grade 3

Exclusion Criteria:

* kidney dysfunction (creatinine >2 mg/dl),
* History of previous liver disease,
* Cardiogenic shock,
* History of myocardial infarction (MI)
* History of coronary artery bypass grafting
* History of allergic response to drugs
* Right ventricular infarction
* Severe hypovolemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoint (whether premature beats,atrial or ventricular tachycardia, atrial or ventricular fibrillation, and atrioventricular block appears;whether severity of chest pain is aggravated,and number of episodes chest pain) | 24hours
  The primary composite endpoint consisted of reperfusion-induced arrhythmia, worsening of chest pain, and no-reflow/slow reflow.
  In perioperative period,we will observe whether the reperfusion-induced arrhythmia including atrial or ventricular premature beats,atrial or ventricular tachycardia, atrial or ventricular fibrillation, and atrioventricular block appears;whether the severity of chest pain is aggravated,and the number of episodes of chest pain will be recorded for patients who complains of chest pain that lasted for at least 30 min within the 24 h following onset of MI;Whether the phenomenon of no-reflow/slow reflow appears.No-reflow and slow flow are diagnosed when the thrombolysis in myocardial infarction(TIMI) flow grade is 2 or lower,despite successful PCI such as balloon angioplasty or stent insertion.

SECONDARY OUTCOMES:
the combined outcome of TIMI frame count (cTFC) of CAG and ST resolution (STR) of ECG | 24hours
  The cTFC was measured according to the method of Gibson et al, to determine blood flow at the time of coronary angiography. The cine frame counts derived from the injection of contrast medium to the peripheral landmark were measured .
  In order to evaluate STR, the total sum of the ST segments elevation from the J point to the point reached 20ms later was calculated from the 12-lead ECG recorded before the start of reperfusion, and 90 min after the completion of reperfusion. The rate of improvement in ST elevation was classified as "complete resolution" (70% or more improvement) and "no resolution" (<70%).

CONTACTS AND LOCATIONS:
Overall Officials: Institute of Cardiovascular Disease Xuzhou Central Hospital, Study Director — Southeast University
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

REFERENCES:
- [Background] Moens AL, Claeys MJ, Timmermans JP, Vrints CJ. Myocardial ischemia/reperfusion-injury, a clinical view on a complex pathophysiological process. Int J Cardiol. 2005 Apr 20;100(2):179-90. doi: 10.1016/j.ijcard.2004.04.013. PMID 15823623
- [Background] Reffelmann T, Kloner RA. The "no-reflow" phenomenon: basic science and clinical correlates. Heart. 2002 Feb;87(2):162-8. doi: 10.1136/heart.87.2.162. No abstract available. PMID 11796561
- [Background] Costantini CO, Stone GW, Mehran R, Aymong E, Grines CL, Cox DA, Stuckey T, Turco M, Gersh BJ, Tcheng JE, Garcia E, Griffin JJ, Guagliumi G, Leon MB, Lansky AJ. Frequency, correlates, and clinical implications of myocardial perfusion after primary angioplasty and stenting, with and without glycoprotein IIb/IIIa inhibition, in acute myocardial infarction. J Am Coll Cardiol. 2004 Jul 21;44(2):305-12. doi: 10.1016/j.jacc.2004.03.058. PMID 15261923
- [Background] Tanaka A, Kawarabayashi T, Nishibori Y, Sano T, Nishida Y, Fukuda D, Shimada K, Yoshikawa J. No-reflow phenomenon and lesion morphology in patients with acute myocardial infarction. Circulation. 2002 May 7;105(18):2148-52. doi: 10.1161/01.cir.0000015697.59592.07. PMID 11994247
- [Background] Limbruno U, De Carlo M, Pistolesi S, Micheli A, Petronio AS, Camacci T, Fontanini G, Balbarini A, Mariani M, De Caterina R. Distal embolization during primary angioplasty: histopathologic features and predictability. Am Heart J. 2005 Jul;150(1):102-8. doi: 10.1016/j.ahj.2005.01.016. PMID 16084155
- [Background] De Luca G, Navarese EP, Suryapranata H. A meta-analytic overview of thrombectomy during primary angioplasty. Int J Cardiol. 2013 Jul 1;166(3):606-12. doi: 10.1016/j.ijcard.2011.11.102. Epub 2012 Jan 28. PMID 22284272
- [Background] Werner GS, Lang K, Kuehnert H, Figulla HR. Intracoronary verapamil for reversal of no-reflow during coronary angioplasty for acute myocardial infarction. Catheter Cardiovasc Interv. 2002 Dec;57(4):444-51. doi: 10.1002/ccd.10375. PMID 12455077
- [Background] Marzilli M, Orsini E, Marraccini P, Testa R. Beneficial effects of intracoronary adenosine as an adjunct to primary angioplasty in acute myocardial infarction. Circulation. 2000 May 9;101(18):2154-9. doi: 10.1161/01.cir.101.18.2154. PMID 10801755
- [Background] Taira N. Nicorandil as a hybrid between nitrates and potassium channel activators. Am J Cardiol. 1989 Jun 20;63(21):18J-24J. doi: 10.1016/0002-9149(89)90200-2. PMID 2525320
- [Background] Ota S, Nishikawa H, Takeuchi M, Nakajima K, Nakamura T, Okamoto S, Setsuda M, Makino K, Yamakado T, Nakano T. Impact of nicorandil to prevent reperfusion injury in patients with acute myocardial infarction: Sigmart Multicenter Angioplasty Revascularization Trial (SMART). Circ J. 2006 Sep;70(9):1099-104. doi: 10.1253/circj.70.1099. PMID 16936418
- [Background] Tsubokawa A, Ueda K, Sakamoto H, Iwase T, Tamaki S. Effect of intracoronary nicorandil administration on preventing no-reflow/slow flow phenomenon during rotational atherectomy. Circ J. 2002 Dec;66(12):1119-23. doi: 10.1253/circj.66.1119. PMID 12499617
- [Background] Lim SY, Bae EH, Jeong MH, Kang DG, Lee YS, Kim KH, Lee SH, Yoon KH, Hong SN, Park HW, Hong YJ, Kim JH, Kim W, Ahn YK, Cho JG, Park JC, Kang JC. Effect of combined intracoronary adenosine and nicorandil on no-reflow phenomenon during percutaneous coronary intervention. Circ J. 2004 Oct;68(10):928-32. doi: 10.1253/circj.68.928. PMID 15459466
- [Background] Kitakaze M, Asakura M, Kim J, Shintani Y, Asanuma H, Hamasaki T, Seguchi O, Myoishi M, Minamino T, Ohara T, Nagai Y, Nanto S, Watanabe K, Fukuzawa S, Hirayama A, Nakamura N, Kimura K, Fujii K, Ishihara M, Saito Y, Tomoike H, Kitamura S; J-WIND investigators. Human atrial natriuretic peptide and nicorandil as adjuncts to reperfusion treatment for acute myocardial infarction (J-WIND): two randomised trials. Lancet. 2007 Oct 27;370(9597):1483-93. doi: 10.1016/S0140-6736(07)61634-1. PMID 17964349
- [Derived] Feng C, Liu Y, Wang L, Niu D, Han B. Effects of Early Intracoronary Administration of Nicorandil During Percutaneous Coronary Intervention in Patients With Acute Myocardial Infarction. Heart Lung Circ. 2019 Jun;28(6):858-865. doi: 10.1016/j.hlc.2018.05.097. Epub 2018 May 22. PMID 29891250